CLINICAL TRIAL: NCT07282288
Title: A Randomized Controlled Study on Autologous Cell Injection Into the Ovaries of Patients With Poor Ovarian Response
Brief Title: A RCT Study on Autologous Cell Injection Into the Ovaries of Patients With POR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Ma Caihong, Chief Physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006761-M20250882; BRWEP2024W094090102 (Other Grant/Funding Number: Beijing Research Ward Excellence Program)
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Poor Ovarian Response
Keywords: Poor ovarian response; Premature ovarian insufficiency; autologous fat vascular matrix components; autologous platelet-rich plasma
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP group (Experimental)
  Interventions: Other: PRP injection
- SVF group (Experimental)
  Interventions: Other: SVF injection
- Control Group (No Intervention)

INTERVENTIONS:
Other: PRP injection — Injecting PRP into the ovaries
  Arms: PRP group
Other: SVF injection — Injecting SVF into the ovaries
  Arms: SVF group

SUMMARY:
Poor ovarian response (POR) is a pathological state where the ovaries do not respond well to the stimulation of gonadotropins. It is mainly characterized by a small number of developing follicles, a high cancellation rate of the ovarian stimulation cycle, a low number of retrieved oocytes, and a low clinical pregnancy rate. Premature ovarian insufficiency (POI) is a special type of this condition and is one of the most difficult infertility diseases to treat. The incidence of POR and POI in reproductive-aged women in China is increasing year by year, making them key and challenging issues in reproductive medicine. New local ovarian cell therapy can improve the microenvironment for follicle development, promote the development and ovulation of "dormant" primordial follicles, and improve the quality of oocytes. This study intends to conduct autologous fat vascular matrix components (SVF) or autologous platelet-rich plasma (PRP) local injection therapy for patients with POR and POI, and conduct a prospective exploratory study to evaluate the safety of this clinical technique. Subsequently, a prospective randomized controlled trial will be conducted to evaluate the safety and efficacy of autologous fat vascular matrix components (SVF) or autologous platelet-rich plasma (PRP) local injection therapy in improving ovarian reserve and IVF-ET outcomes. This study is expected to improve the fertility of patients with POR from the perspective of autologous cell therapy. The autologous SVF and PRP local injection techniques do not involve ethical barriers, are easy to standardize the diagnosis and treatment process and operation system, and are suitable for clinical translation and promotion.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have fertility requirements and are seeking IVF treatment
2. Age ≤ 45 years old, infertility duration ≥ 1 year
3. Meeting the diagnostic criteria for POI or the Poseidon diagnostic criteria for POR
4. Previous controlled ovarian stimulation resulted in no more than 3 oocytes retrieved and/or no transplantable embryos and/or previous embryo implantation failure ≥ 2 times
5. Uterus and bilateral adnexa are intact
6. BMI 22 - 29 kg/m²
7. Participants must have given informed consent for this study and voluntarily signed a written informed consent form.

Exclusion Criteria:

1. Congenital abnormalities of reproductive organs
2. Septicemia, platelet dysfunction syndrome and severe thrombocytopenia and other coagulation disorders or other hematological diseases
3. Suffering from autoimmune diseases or other endocrine disorders, with abnormal thyroid function and uncontrolled condition
4. Having a mass in the adnexal area with an unclear benign or malignant nature
5. Complicated with severe cardiovascular and cerebrovascular diseases, malignant tumors, hematological diseases and mental disorders, patients with impaired function of important organs
6. Those who have used systemic corticosteroids within the last 2 weeks, or used antiplatelet drugs such as aspirin within the last 48 hours
7. In the acute inflammatory stage
8. Those with a history of venous thrombosis or pulmonary embolism during the screening period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved oocytes | 6month

SECONDARY OUTCOMES:
anti-Müllerian hormone level | 6 month
Number of antral follicles | 6 month
clinical pregnancy rate | 1 year